CLINICAL TRIAL: NCT07050433
Title: PCF Challenge 2023 Correlate Biomarkers for the SYNERGY- 201 Study
Brief Title: Correlate Biomarkers for the SYNERGY- 201 Study
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00115687
Record Dates: First submitted 2025-06-04; First posted 2025-07-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; SYNERGY-201; SX-682; CXCR2 inhibition
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Men who are participating in the SYNERGY-201 clinical trial (NCT06228053).: Men with metastatic castration resistant prostate cancer (mCRPC) who are participating in the SYNERGY-201 clinical trial (NCT06228053) and who also agree to participate in this study will have blood collected for circulating tumor DNA (ctDNA) and immune cell profiling assessments and other research assessments at baseline, Cycle 3 Day 1 of SYNERGY-201 and at the time of the decision to discontinue the SYNERGY-201 study drug. A subset of up to 20 participants will also undergo tumor biopsies at the baseline and Cycle 3 Day 1 visits of SYNERGY-201.
  Interventions: Diagnostic Test: CXCR2 as a biomarker

INTERVENTIONS:
Diagnostic Test: CXCR2 as a biomarker — CXCR2 biomarker expression will be measured in tumor and immune cell samples

SUMMARY:
This study is a companion to the SYNERGY-201 clinical trial (NCT06228053), which investigates SX-682 and enzalutamide in individuals with prostate cancer. Individuals must be participating in SYNERGY-201 in order to participate in this study. The purpose of this companion study is to learn more about biomarkers, particularly a biomarker called CXCR2, and investigate if CXCR2 can predict who will receive benefit from the SYNERGY-201 drug combination. This study will also investigate how CXCR2 and other biomarkers change over time when participants receive the SYNERGY-201 drug combination. CXCR2 is of particular interest because the SYNERGY-201 drug, SX-682, inhibits CXCR2. After participants provide consent, blood samples will be collected for research purposes at three SYNERGY-201 visits (Baseline, Cycle 3 Day 1 and End of Study Drug). Up to 20 participants will also receive tumor biopsies at the Baseline and SYNERGY-201 Cycle 3 Day 1 visits. Clinical and study data collected as part of SYNERGY-201 will also be used for this study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for this study and HIPAA authorization for the release of personal health information.
* Age >18
* Participating in the SYNGERY-201 clinical trial.

Exclusion Criteria:

* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study
* History or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the subject's participation for the full duration of the study
* History or current evidence of any condition, therapy, or laboratory abnormality that is not in the best interest of the subject to participate (in the opinion of the treating investigator)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes men with metastatic castration resistant prostate cancer (mCRPC) who are participating in the SYNERGY-201 clinical trial as defined in the eligibility criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Tumor CXCR2 biomarker expression associated with clinical benefit (CB) | 6 months from Cycle 1 Day 1 (each cycle is 21 days)
  The association between tumor CXCR2 (dichotomized as absent or present CXCR2 levels in tumor at baseline as compared to negative control tissue) and CB will be measured using an odds ratio with 95% CI.
Number of participants with Immune cell CXCR2 biomarker expression associated with clinical benefit (CB) | 6 months from Cycle 1 Day 1 (each cycle is 21 days)
  The association between immune cell CXCR2 (dichotomized as present or absent in any myeloid immune cell subset) and CB will be measured using an odds ratio with 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No